CLINICAL TRIAL: NCT06696495
Title: Evaluation of Morphofunctional and Baropodometric Changes in the Foot and Ankle of Pregnant Women: Longitudinal Study from the Pregestational Stage to the Postpartum Period
Brief Title: Evaluation of Morphofunctional and Baropodometric Changes in Pregnant Women
Acronym: FOOTpreg
Status: Not yet recruiting | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, ANA MARIA RAYO PEREZ, Principal Investigator, University of Seville
Other Study IDs: FOOTPREGNANT
Record Dates: First submitted 2024-10-31; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy Related; Foot Diseases
Keywords: pregnancy; foot diseases; Postural Balance; Foot Morphology
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnancy women: Each participant will undergo various tests to assess morphofunctional and baropodometric changes in the foot and ankle. These tests will include measuring the size and width of the foot using a 3D scanner, assessing the height of the plantar arch using a podoscope, and applying functional scales such as the AOFAS (Ankle and Foot Outcome Score), the FPI (Foot Posture Index) and the FFI (Foot Function Index). In addition, plantar pressure distribution and centre of pressure (COP) will be analysed to identify variations in stability and balance during pregnancy.
  Interventions: Diagnostic Test: Measurement of the size and width of the foot

INTERVENTIONS:
Diagnostic Test: Measurement of the size and width of the foot — Assessment of the height of the plantar arch using a podoscope, and application of functional scales such as the AOFAS (Ankle and Foot Outcome Score), the FPI (Foot Posture Index) and the FFI (Foot Function Index). In addition, the distribution of plantar pressure and the centre of pressure (COP)

SUMMARY:
Pregnancy causes physiological and biomechanical changes in the female body, such as weight gain and hormonal changes, which can affect the structure and function of the foot and ankle. These adaptations can influence gait, balance and stability. However, the temporal evolution of these changes in the foot and ankle before, during and after pregnancy is not well documented. This study aims to characterize and quantify these changes, as well as their impact on foot function, with the aim of contributing to the prevention and management of podiatric and orthopedic problems in pregnant women.

DETAILED DESCRIPTION:
Pregnancy causes physiological and biomechanical changes in the female body, such as weight gain and hormonal changes, which can affect the structure and function of the foot and ankle. These adaptations can influence gait, balance and stability. However, the temporal evolution of these changes in the foot and ankle before, during and after pregnancy is not well documented. This study aims to characterize and quantify these changes, as well as evaluate their impact on foot function, thus contributing to the prevention and management of podiatric and orthopedic problems in pregnant women.

The general objective of this study is to evaluate the morphofunctional and baropodometric changes of the foot and ankle in pregnant women from the pre-gestational period to the postpartum period. Specific objectives include determining changes in foot and ankle size and width at different stages, assessing foot function using the AOFAS (Ankle and Foot Outcome Score), FPI (Foot Posture Index) and FFI (Foot Function Index) indices, analyzing plantar pressure distribution and baropodometric changes, and correlating morphofunctional and baropodometric changes with weeks of gestation and maternal weight.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women between 20 and 35 years old.
2. If pregnant, they must be in the first trimester of pregnancy (before week 12).
3. Absence of chronic or acute pathologies that may interfere with the analysis of biomechanical variables (arthritis, vascular or metabolic problems).
4. Not having had previous foot or ankle surgeries.

Exclusion Criteria:

1. Women with multiple pregnancies (twin or multiple pregnancies increase biomechanical variations).
2. Conditions that affect gait or foot structure (arthritis, neuropathies, or other orthopedic problems).
3. History of previous foot or ankle injuries that may alter measurements.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The objective is to know the morphofunctional changes of the foot during pregnancy
Study Population: The study population will be composed of healthy women between 20 and 35 years of age who meet the established inclusion criteria. If the participants are pregnant, they must be in the first trimester of pregnancy, that is, before week 12. It will be ensured that they do not have chronic or acute pathologies, such as arthritis or vascular or metabolic problems, that could interfere with the analysis of the biomechanical variables. In addition, the participants must not have had previous surgeries on the foot or ankle. On the other hand, women with multiple pregnancies will be excluded from the study, as well as those who suffer from conditions that affect the gait or the structure of the foot, and those who have a history of previous injuries to the foot or ankle that could alter the measurements.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Ankle and Foot Outcome Score | 3 times. before pregnancy, at 4 months of pregnancy and at 3 months post-pregnancy
  Completion of the scale before pregnancy, at 4 months of pregnancy and at 3 months post-pregnancy. The score is 0 to 100 points.
Foot Fuction Index Score | 3 times. Before pregnancy, at 4 months of pregnancy and at 3 months post-pregnancy
  Completion of the scale before pregnancy, at 4 months of pregnancy and at 3 months post-pregnancy. The score is 0 to 100 points.
Measurement of the length and width of the foot | 3 times. Before pregnancy, at 4 months of pregnancy and at 3 months post-pregnancy
  Completion of the scale before pregnancy, at 4 months of pregnancy and at 3 months post-pregnancy

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clinica Rayo, Seville, SEVILLA
  - Universidad de Sevilla, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: No